CLINICAL TRIAL: NCT05128357
Title: IMPACT_BD (IMProving AdherenCe to Treatment in Behçet's Disease)
Acronym: IMPACT_BD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Rosaria Talarico, MD, PhD, Azienda Ospedaliero, Universitaria Pisana
Other Study IDs: RTalarico
Record Dates: First submitted 2021-11-09; First posted 2021-11-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Behçet Disease
Keywords: Behçet; adherence to treatment; multistakeholder approach
MeSH Terms: conditions — Behcet Syndrome; Treatment Adherence and Compliance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: the study is observational, no intervention foreseen — the study does not foresees any intervention, since it is a multi step observational study.

SUMMARY:
Behçet's disease (BD) is an autoimmune, rare, and severe multisystemic inflammatory disease characterized by recurrent oral aphthous ulcers, genital ulcers, skin lesions, and both anterior and posterior uveitis; articular, vascular, gastroenteric and neurological involvement may also occur. The multi-organ involvement and the wide range of clinical spectrum make the diagnosis of BD challenging. Adherence has been defined as the "extent to which a person's behavior (in terms of taking medications, following diets, or executing other lifestyle changes) corresponds with agreed recommendations from a health care provider". The lack of medication adherence leads to poorer health outcomes for the patients, which affect quality of life, generate economic loss for the healthcare system and trigger uncertainty for the healthcare prescribers in dealing with the disease treatment. This challenge is particularly important in BD. The present study is therefore aimed at exploring the main reasons for low- or non-adherence to treatments in BD and to create a specific tool able to catch and monitor the reasons for low- or non-adherence in BD over time.

Objectives

* to explore the unmet needs in treatment adherence
* to create a toll aimed at identifying and monitoring the reasons of low treatment adherence
* to plan specific actions aimed at improving treatment adherence in BD

DETAILED DESCRIPTION:
Methodology The methodology includes 5 consequent phases, summarized below. Phase A. Panel creation - The first step foresees the creation of a multi-stakeholder panel, that will include clinicians, BD patients' representatives, BD caregiver' representatives and other experts (economists, psychologist, pharmacists, etc). The multi-stakeholder approach will contribute to improve the identification of the different barriers, perspectives and unmet needs of the different stakeholders and to identify the patients' outcomes to be included in the tool. The panel will be created by launching an international call for interest.

Phase B. Co-design process - An ad hoc survey will be created in co-design with the different stakeholders in order to capture all the different dimensions, barriers and needs that are involved in the process of treatment adherence, as well to ensure the accessibility and understandability of the survey. The survey will include two main sections: one section with questions and a section dedicated to narrative medicine, that will provide a limited space for patients and caregivers to express their perspective, views, needs and priorities in terms of treatment adherence.

The survey will be translated in different languages to ensure a wide dissemination across different countries.

Phase C. Launch of the survey - This phase foresees the upload of the survey into the EU Survey and the launch of the survey across the different centers involved in the study.

BD patients and caregivers will be able to access the survey online for at least 3 months in order to reach the greatest number possible of respondents.

Phase D. Data analysis, workshop and agreement - The answers to the questions and the contributions provided in the narrative medicine section will be elaborated in order to identify the main barriers and unmet needs related to treatment adherence in BD patients and caregivers.

In addition, an online workshop will be organized in order to:

* elaborate and discuss the results of the survey;
* co-design and reach a formal agreement on the tool that will enable the identification and the monitoring of BD treatment adherence during the clinical follow-up of BD patients.

Phase E. Pilot phase for validation - The final tool will then be translated in different languages and will be adopted in a pilot phase that will involve at least 300 BD patients and caregivers form different countries. The results of the pilot phase will be discussed in the panel described in Phase A and the tool will be refined according to the results gathered in the pilot. The final tool will then be published in a scientific paper and distributed to BD experts and patients' organisations for adoption. In addition, based on the results of the pilot phase, a list of future actions aimed at improving treatment adherence in BD patients will be produced with the support of members of the co-design panel organized in Phase A.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Behçet's disease

Exclusion Criteria:

* BD patients < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At leads 300 patients with a diagnosis of Behçet's disease
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-11-16 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
To explore the unmet needs in treatment adherence in Behçet's disease patients | From November 2021 to middle May 2022
  An ad hoc survey will be created in co-design with the different stakeholders in order to capture all the different dimensions, barriers and needs that are involved in the process of treatment adherence, as well to ensure the accessibility and understandability of the survey. The answers to the questions and the contributions provided in the narrative medicine section will be elaborated in order to identify the main barriers and unmet needs related to treatment adherence in BD patients and caregivers.
The creation of a co-designed tool aimed at assessing the causes and barriers of low- or non adherence in BD patients; | From May 2022 to July 2022
  he final tool will then be translated in different languages and will be adopted in a pilot phase that will involve at least 300 BD patients and caregivers form different countries. The results of the pilot phase will be discussed in the panel described in Phase A and the tool will be refined according to the results gathered in the pilot.

CONTACTS AND LOCATIONS:
Locations (1):
- AOUPisana, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Talarico R, Marinello D, Manzo A, Cannizzo S, Palla I, Ticciati S, Gaglioti A, Trieste L, Pisa L, Badalamenti L, Randisi G, Del Bianco A, Lorenzoni V, Turchetti G, Mosca M. Being a caregiver of a Behcet's syndrome patient: challenges and perspectives during a complex journey. Orphanet J Rare Dis. 2021 Oct 18;16(1):436. doi: 10.1186/s13023-021-02070-2. PMID 34663419
- [Result] Pirri S, Marinello D, Lorenzoni V, Andreozzi G, Bazzani A, Del Bianco A, Turchetti G, Mosca M, Talarico R. Adherence to treatment in Behcet's syndrome: a multi-faceted issue. Clin Exp Rheumatol. 2021 Sep-Oct;39 Suppl 132(5):88-93. doi: 10.55563/clinexprheumatol/1lx7a5. Epub 2021 Sep 30. PMID 34596034